CLINICAL TRIAL: NCT04615741
Title: Improving Health and Wellness During COVID-19
Brief Title: Finding Wellness in the Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Responsible Party: Principal Investigator, Cheryl Currie, Associate Professor, University of Lethbridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-096
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Wellness 1; Addiction; Stress, Psychological; Covid19
MeSH Terms: conditions — Behavior, Addictive; Stress, Psychological; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trauma Informed Yoga (Experimental): Participants will receive 8 x 60 min group-based yoga sessions, delivered synchronously over Zoom.
  Interventions: Behavioral: Trauma Informed Yoga
- Trauma Informed Psychotherapy (Experimental): Participants will receive 8 x 90 min group-based psychotherapy sessions, delivered synchronously over Zoom.
  Interventions: Behavioral: Trauma Informed Psychotherapy
- Control (No Intervention): These participants will not receive an intervention.

INTERVENTIONS:
Behavioral: Trauma Informed Yoga — One licensed yoga instructor, trained in trauma-informed yoga delivery, will lead the online sessions. Participants will be instructed to engage in the class from a mat or chair in their home or move between them as the class unfolds. The instructor will begin the class by introducing the week's theme (e.g. grounding and safety, non-attachment, imprints of the past and impacts on our reactions to COVID-19, connection to nature), followed by a breath practice (10 min), a yoga practice (50 min), a meditation practice (10 min), and closing words (10 min).
  Arms: Trauma Informed Yoga
Behavioral: Trauma Informed Psychotherapy — Two licensed counsellors (MSW-trained) will co-facilitate the online version of this program. Facilitators will begin the session by introducing the week's theme (e.g. setting goals while working from home, being mindful, health coping) (10 min), followed by a lecture and activity to integrate learning (e.g. large and small group discussion using Zoom break out rooms, journaling) (70 min), and closing words (10 min).
  Arms: Trauma Informed Psychotherapy

SUMMARY:
There is an immediate need for population-level intervention research to address the impacts of the coronavirus disease 2019 (COVID-19) pandemic and its containment measures on mental health and substance use (MHSU). While online programs are available to address these issues, they are often delivered in an asynchronous format with relatively low therapist or health coaching guidance. As highlighted by a recent systematic review, positive outcomes for online mental health programs are tied to the intensity of therapist or coaching guidance, which increases cost and reduces population access to more effective online options. A way to offset cost while maintaining effectiveness is to offer MHSU programs to groups online, rather than individually. In 2019, the investigators launched an RCT to test gender-stratified group interventions to address MHSU among community-based Indigenous and non-Indigenous adults in southern Alberta. The investigators implemented the interventions with more than 200 adults before the study was paused due to COVID-19.

DETAILED DESCRIPTION:
The primary objective of this project is to adapt two existing mental health and substance use interventions and RCT for online delivery, COVID-19 impacts, and province-wide spread. The second objective is to test if an online group body-oriented intervention (trauma-sensitive yoga) that has been designed to increase awareness of physical sensations, is superior to an online group verbal narrative intervention (mental wellness talking circle), and to control group. The investigators theorize that the body-oriented intervention may offer the opportunity to reprogram automatic physiologic hyperarousal in response to COVID-19 triggers and increase positive body awareness, and mindful attention to the ways in which habitual self-protective behaviours like substance use may be impacting health. The third objective is to examine the impacts of the interventions on adults with pre-existing MHSU issues, and those with previous experiences that may make them more susceptible to MHSU problems during COVID-19. The investigators will track other supports the participants engage during the study and the perceived impacts of these supports on the outcomes with the goal of shedding light on how to best match COVID-19 related services to adults who need them the most.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-75 years living in Alberta, Canada
* Need to have reliable access to the internet, a device with a webcam for the next 2 months
* Need to self-identify that they are currently struggling with at least one of: stress eating, alcohol use, drug use, tobacco use, or gambling during the pandemic

Exclusion Criteria:

* Non-community dwelling
* Do not currently reside within Alberta, Canada

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Changes in Tobacco Use | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Participants will be asked to self-report if tobacco use has changed during the pandemic via a 5-point likert. Options range from increased a lot to decreased a lot. If participants indicate their tobacco use has changed, they will be asked to identify the primary reason for this change. Changes in tobacco use will be re-assessed at each time point.
Changes in Alcohol Use | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Past year alcohol consumption will be assessed through the Alcohol Use Disorder Identification Test (AUDIT). Scores on the AUDIT range from 0 to 40; a score over 8 is indicative of problematic or hazardous alcohol use. Changes in alcohol consumption since the beginning of the pandemic will be identified through a 5-point likert. Changes in alcohol use will be re-assessed at each time point.
Changes in Drug Use | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Past year drug use will be assessed through the Drug Use Disorders Identification Test (DUDIT). Possible scores on the DUDIT range from 0 to 44; scores greater than 2 or 6 are indicative of risky or harmful drug habits for women and men, respectively. A score of 25 or more suggests the individual is probably heavily dependent on drugs. Participants will also be asked to identify which drugs they currently use, the main reasons for using drugs, and whether their drug use has changed during the pandemic. Changes in drug use will be re-assessed at each time point.
Changes in Gambling | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Gambling will be assessed via the 9-item Problem Gambling Severity Index (PGSI). The items are measured on a 5-point likert with frequencies from "less than once a month" to "daily or almost daily". A cut-score ≥5 will be used (lower scores indicative of non-problem gambling); the PGSI has a high internal consistency (α = 0.86) and is considered the measure of choice for non-clinical use.
Changes in Post-Traumatic Stress Symptoms | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  A revised version of the Primary Care - Post Traumatic Stress Disorder - 5 (PC-PTSD-5) scale will be assessed to determine experiences of trauma in relation to COVID-19. The scale was revised to specifically ask about COVID-19. Scores range from 0 (no risk) to 5 (high risk). A cut-score of 3 will be used to differentiate high- and low-risk scores. The PC-PTSD has good sensitivity (r = 0.78) and sensitivity (r = 0.87).
Changes in Depression Symptoms | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Depression will be screened using the 10-item Centre for Epidemiological Studies Depression Scale (CES-D-10). The CES-D-10 is a short self-report scale to measure depressive symptoms in a general population. Psychometric evaluation has shown the CES-D-10 to have high internal consistency, though with variability across populations (Cronbach's α = 0.71 to 0.90) and good construct validity (r = 0.78).
Changes in Anxiety Symptoms | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  The 6-item State-Trait Anxiety Inventory (STAI-6) will be used to measure anxiety reflective of both adverse situations (state anxiety) and personality traits associated with higher levels of anxiety (trait anxiety). STAI-6 produces scores like its longer 20-item version, showing good reliability (Cronbach's α = 0.82) with sensitivity to differing degrees of anxiety. Possible scores range from 20 to 80; "normal scores" range from 34 to 36. Higher scores represent higher amount of anxiety.

SECONDARY OUTCOMES:
Changes in Eating Behaviour | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Changes in eating behaviours will be assessed by questions asking if food consumption and unhealthy food consumption have changed since the onset of the pandemic via a 5-point likert scale (increased a lot to decreased a lot). If participants indicate they have changed their food consumption, a qualitative question will ask them to describe why they think their behaviour has changed.
Changes in Sleeping Behaviour | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Participants will be asked to rate how the quantity and quality of their sleep has changed since the pandemic started via 5-point likert scales (increased a lot to decreased a lot).
Changes in Physical Activity | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Physical activity will be assessed through the International Physical Activity Questionnaire - Short Form. The questionnaire asks about frequency and duration of vigorous (VPA) and moderate physical activity (MPA) over the past 7 days. Weekly Metabolic Equivalents (MET) minutes will be calculated based on responses. Participants will be categorized into high (>1500 MET min/week with 3+ days of VPA or >3000 METmin/week with 7+ days of MVPA); medium (5+ days of 20+ minutes of VPA per day, 5+ days with 30+ minutes of MPA per day, or 5+ days of MVPA that achieves 600+ MET min/week); low (participant does not meet other cut points).
  Frequency and duration of walking and sitting time are also assessed. The IPAQ has good reliability and criterion validity. Participants will also be asked if their PA and sedentary behaviour levels have changed during the pandemic (5-point likert; options: increased a lot to decreased a lot).
Changes in Resilience | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  The 10-item Connor-Davidson Resilience Scale (CD-RISC 10) is a widely used measure to assess self-perceived resilience. Evaluations of the CD-RISC 10 have shown good internal consistency (Cronbach's α = 0.85), a strong positive association with the longer 25-item CD-RISC (r = 0.92). Scores range from 0 to 40; a higher score is indicative of higher resilience.
Changes in Self-Esteem | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Self-esteem will be measured using the 10-item Rosenberg Self Esteem Scale. The scale is a widely used measure that correlates well with other measures of self-esteem and has strong internal consistency (0.92) and test-retest reliability (0.88). Scores range from 4 to 40; a higher score indicates higher self esteem. Participants will also be asked how their self-esteem has changed since the beginning of the pandemic.
Changes in Loneliness | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Loneliness will be evaluated using a shortened (3 item) version of the UCLA Loneliness Scale. This scale asks about feelings of companionship, being left out, and being isolated from others in the last month, with a 3-item list of answer options (hardly ever, some of the time, often). This scale has good reliability (r = 0.73), validity, and internal consistency (Cronbach's α = 0.84-0.94). The scale also showed convergent validity with other commonly used measures of loneliness. Scores range from 1 to 9; higher scores indicate higher levels of loneliness.
Changes in Dissociative Experiences | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  The Brief Dissociative Experiences Scale is an 8-item tool that assesses the severity of dissociative experiences in adults. The scale items are summed and averaged to describe the severity of dissociative experiences as none (0), mild (1), moderate (2), severe (3), or extreme (4). The brief scale was found to be reliable, easy to use, and clinically useful in the DSM-5 Field Trials. Scores range from 0 to 32; a higher score indicates a greater severity of dissociative experiences.

OTHER OUTCOMES:
Changes in Coping Strategies | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Coping strategies and perceived ability to cope during the pandemic will be assessed through four self-reported questions. Participants will be asked how well they are coping with the pandemic on a 5-point likert, options will range from 'excellent' to 'poor'. Participants will be asked to identify things that are helping them to cope from a list of 18 items. Current life satisfaction will be assessed with a single question with options ranging from "very satisfied" to "very dissatisfied". Participants will also be asked to identify up to 3 things they wish they could change right now in their life.
Changes in Relationships and Belonging | Baseline, Mid-point (4-weeks), Post-intervention (8-weeks), 3-month Follow Up
  Participants will be asked to self-report feelings of belonging to their local and work communities. They will also be asked to self-report changes to the quality or stress associated with their romantic relationships and the presence of abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Currie, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- University of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data relevant to the researcher's research question may be shared upon a reasonable request
Time Frame: After April 2021, for up to 10 years
Access Criteria: Researchers must make a reasonable request to the PI